CLINICAL TRIAL: NCT04750473
Title: Phase 1 Feasibility Trial: Improved Staging of Lobular Breast Cancer With Novel Amino Acid Metabolic and Tumor Neovasculature Receptor Imaging
Brief Title: Fluciclovine and PSMA PET/CT for the Classification and Improved Staging of Invasive Lobular Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, David M Schuster, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00000675; NCI-2020-00366 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); WINSHIP4933-19 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2021-02-09; First posted 2021-02-11 (Actual); Results first posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Invasive Breast Lobular Carcinoma; Metastatic Breast Lobular Carcinoma; Prognostic Stage IV Breast Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Lobular | interventions — fluciclovine F-18; gallium 68 PSMA-11; 68Ga-DKFZ-PSMA-11; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (Ga PSMA, fluciclovine F18, PET/CT) (Experimental): Patients receive gallium Ga 68-labeled PSMA-11 IV and undergo a PET/CT scan over 30 minutes. On a separate day, patients receive fluciclovine F18 IV and undergo a PET/CT scan over 30 minutes.
  Interventions: Procedure: Computed Tomography; Drug: Fluciclovine F18; Drug: Gallium Ga 68 Gozetotide; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT scan
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Drug: Fluciclovine F18 — Given IV
  Other Names: (18F)Fluciclovine; (18F)GE-148; 18F-Fluciclovine; [18F]FACBC; Anti-(18f)FABC; Anti-1-Amino-3-[18F]Fluorocyclobutane-1-Carboxylic Acid; Anti-[18F] FACBC; Axumin; Fluciclovine (18F); FLUCICLOVINE F-18; GE-148 (18F); GE-148 F-18
Drug: Gallium Ga 68 Gozetotide — Given IV
  Other Names: (68)Ga labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; (68)Ga-labeled Glu-urea-Lys(Ahx)-HBED-CC; (68)Ga-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68)Gallium-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68Ga)Glu-urea-Lys(Ahx)-HBED-CC; 68Ga-DKFZ-PSMA-11; 68Ga-HBED-CC-PSMA; 68Ga-labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; 68Ga-PSMA; 68Ga-PSMA-11; 68Ga-PSMA-HBED-CC; [68Ga] Prostate-specific Membrane Antigen 11; [68Ga]GaPSMA-11; Ga PSMA; Ga-68 labeled DKFZ-PSMA-11; Ga-68 labeled PSMA-11; GA-68 PSMA-11; Gallium Ga 68 PSMA-11; Gallium Ga 68-labeled PSMA-11; GALLIUM GA-68 GOZETOTIDE; Gallium-68 PSMA; Gallium-68 PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; GaPSMA; PSMA-HBED-CC GA-68
Procedure: Positron Emission Tomography — Undergo PET/CT scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This phase I trial studies how well fluciclovine positron emission tomography (PET)/computed tomography (CT) and PSMA PET/CT work in helping doctors understand and classify invasive lobular breast cancer in patients with invasive lobular breast cancer that is suspicious for or has spread to other places in the body (metastasized). Fluciclovine and PSMA are radiotracers used in PET/CT imaging scans that emit radiation. The PET/CT scan than picks up the radiation being released to create a picture from within the body. Information learned from this study may help researchers learn how to better identify metastatic disease in invasive lobular breast cancer patients which will impact appropriate staging.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Improve detection of metastasis with fluciclovine F18 (fluciclovine) and gallium Ga 68-labeled PSMA-11 (PSMA) PET versus best standard of care conventional imaging, as confirmed with histology.

II. Determine concordance and discordance of invasive lobular breast cancer (ILC) detection with PSMA versus fluciclovine PET, as confirmed with histology.

EXPLORATORY OBJECTIVE:

I. Establish the role of circulating tumor deoxyribonucleic acid (DNA) (ctDNA) directed to ESR1 and PI3K DNA in characterizing the degree of tumor burden as identified by metabolic amino acid transport and tumor neovasculature receptor imaging.

OUTLINE:

Patients receive gallium Ga 68-labeled PSMA-11 intravenously (IV) and undergo a PET/computed tomography (CT) scan over 30 minutes. On a separate day, patients receive fluciclovine F18 IV and undergo a PET/CT scan over 30 minutes.

After completion of study, patients are followed up in 5-10 business days, and then up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Treatment naive biopsy proven ILC patients with ILC
* Either: a) clinical or imaging suspicion of metastatic disease; or b) proven metastatic disease but in whom there is suspicion of an even greater tumor burden that could change therapy approach
* Ability and willingness to undergo biopsy if needed per standard of care for possible metastasis which could change therapy approach

Exclusion Criteria:

* Pregnancy. Qualitative or quantitative serum or urine pregnancy test will be done in women of childbearing potential within 24 hours before PET

  * A female of childbearing potential (FCBP) is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 12 consecutive months (if age > 55 years); if the female subject is < 55 years and she has been naturally postmenopausal for > 1 year her reproductive status has to be verified by additional lab tests (< 20 estradiol OR estradiol < 40 with follicle-stimulating hormone [FSH] > 40 in women not on estrogen replacement therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-07-16 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2024-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Schuster, MD, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Mushtaq A, Lawal IO, Muzahir S, Friend SC, Bhave M, Meisel JL, Torres MA, Styblo TM, Graham CL, Kalinsky K, Switchenko J, Ulaner GA, Schuster DM. Prospective investigation of amino acid transport and PSMA-targeted positron emission tomography for metastatic lobular breast carcinoma. Eur J Nucl Med Mol Imaging. 2024 Nov;51(13):4073-4082. doi: 10.1007/s00259-024-06830-7. Epub 2024 Jul 8. PMID 38976035

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diagnostic (Ga PSMA, Fluciclovine F18, PET/CT)
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (Ga PSMA, Fluciclovine F18, PET/CT)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Verified Detection Rate for Metastasis
Description: Detection rates are compared between fluciclovine positron emission tomography (PET) and conventional imaging. Paired detection rates will be assessed using McNemar's test. Detection rates will be reported for each method, and 95% confidence intervals will be estimated using the Clopper-Pearson approach. Rates of concordant/discordant observations will be reported.
Time Frame: Up to 105 days
Measure: Mean (95% Confidence Interval); unit: SUVMax
Groups:
- F-Fluciclovine; Ga-PSMA-11: Patients receive gallium Ga 68-labeled PSMA-11 IV and undergo a PET/CT scan over 30 minutes. On a separate day, patients receive fluciclovine F18 IV and undergo a PET/CT scan over 30 minutes.
  Computed Tomography: Undergo PET/CT scan
  Fluciclovine F18: Given IV
  Gallium Ga 68 Gozetotide: Given IV
  Positron Emission Tomography: Undergo PET/CT scan
Arm/Group | F-Fluciclovine | Ga-PSMA-11
Number analyzed (Participants) | 20 | 20
SUVMax | 5.9 [3 to 8.8] | 5.5 [0.3 to 10.7]

2. Primary Outcome: Verified Detection Rate for Invasive Lobular Breast Cancer
Description: Compared between gallium Ga 68-labeled PSMA-11 PET, fluciclovine PET, and conventional imaging. Paired detection rates will be assessed using McNemar's test. Detection rates will be reported for each method, and 95% confidence intervals will be estimated using the Clopper-Pearson approach. Rates of concordant/discordant observations will be reported.
Time Frame: Up to 105 days
Measure: Mean (95% Confidence Interval); unit: SUVMax
Arm/Group | F-Fluciclovine | Ga-PSMA-11
Number analyzed (Participants) | 20 | 20
SUVMax | 7.8 [5.1 to 10.5] | 4.6 [2.9 to 6.3]

ADVERSE EVENTS:
Time Frame: Up to 45 days
Description: CTAE v5
Arm/Group | Diagnostic (Ga PSMA, Fluciclovine F18, PET/CT)
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-29): https://cdn.clinicaltrials.gov/large-docs/73/NCT04750473/Prot_SAP_001.pdf
  • Informed Consent Form (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/73/NCT04750473/ICF_000.pdf